CLINICAL TRIAL: NCT05567627
Title: Single Arm, Multicenter, Open and Dose-escalation Clinical Study on Safety, Tolerance, and Efficacy of GC301, an AAV-Delivered Gene Transfer Therapy in Patients With Infantile-onset Pompe Disease
Brief Title: Clinical Exploration of Adeno-associated Virus (AAV) Expressing Human Acid Alpha- Glucosidase (GAA) Gene Therapy for Patients With Infantile-onset Pompe Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seventh Medical Center of PLA General Hospital (Other)
Collaborators: GeneCradle Therapeutics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC301-IOPD-003
Record Dates: First submitted 2022-09-25; First posted 2022-10-05 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Infantile-onset Pompe Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Initial dose cohort (Experimental): 1.2x10^14 vg/kg of GC301 administered via intravenous infusion
  Interventions: Biological: Genetic: GC301

INTERVENTIONS:
Biological: Genetic: GC301 — GC301, is an adeno-associated virus 9 (AAV9) vector delivering a functional copy of the human GAA gene

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of GC301 adeno-associated virus vector expressing codon-optimized human acid alpha-glucosidase (GAA) as potential gene therapy for Pompe disease. Patients diagnosed with infantile-onset Pompe disease who are younger than 6 months old will be studied.

ELIGIBILITY:
Inclusion Criteria:

* The patient's legal guardian(s) must be able to understand the purpose and risks of the study and voluntarily provide signed and dated informed consent prior to any study-related procedures being performed;
* The patient must be no older than 6 months;
* The patient must be diagnosed with infantile-onset Pompe disease.

Exclusion Criteria:

* Class IV patient based on Modified Ross Heart Failure Classification for Children;
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3x upper limit of normal (ULN), alkaline phosphatase (ALP) > 2x ULN (with the exception of liver abnormalities related to Pompe disease);
* Patient has severe organ dysfunction, such as liver and kidney failure (Liver failure: patients may have liver failure syndrome, including fatigue, severe gastrointestinal symptoms; clinical examination found prolonged prothrombin time, prothrombin activity less than 40%; Neuropsychiatric symptoms, such as restlessness, changes in personality and behavior, lethargy, coma, etc.; Toxic tympanic bowel, ascites, multiple organ dysfunction, etc.; hyperalbuminemia exceeding 171 μmol/L, hypoalbuminemia. Renal failure: creatinine exceeding 110 μmol/L, or glomerular filtration rate less than 100 mL/min), congenital/acquired encephalopathy, etc.;
* Patient with congenital organ absence;
* Patient with primary immunodeficiency;
* Patient who is positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis C antibody, or treponema pallidum antibody;
* Patient with a history of glucocorticoid allergy；
* Patient who has participated in a previous gene therapy research trial;
* Patient who has any concurrent clinically significant major disease or any other condition that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability over time | Infusion to the end of study, average 1 year
  Frequency of adverse events (AEs), serious adverse events (SAEs), and changes from baseline in relevant clinical laboratory tests

SECONDARY OUTCOMES:
Proportion of patients treated w/ GC301 who were alive and free of ventilator support at 12 months of age; | 52 weeks
Changes from baseline Left Ventricular Mass (LVM) | 26 and 52 weeks
Changes from baseline creatine kinase (CK) | 26 and 52 weeks

OTHER OUTCOMES:
Change from baseline glycogen content in muscle tissue | 26 and 52 weeks
Change from baseline acid alpha-glucosidase (GAA) enzyme in muscle and blood | 26 and 52 weeks
Improvement in patient's motor function | 52 weeks
  To evaluate the changes in patient's mobility and physical ability using Hammersmith Infant Neurological Examination (HINE) scores
The viral load of adeno-associated virus (AAV) vector | At multiple time points from pre-dose through up to 1 years post-dose
  To assess the change of AAV vector copy numbers within 52 weeks after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayi Children's Hospital, Seventh Medical Center, PLA general hospital, Beijing, Beijing Municipality, China